CLINICAL TRIAL: NCT04326049
Title: Performance of Large Loop Excision of the Transformation Zone Using Videocolposcopy Versus Binocular Colposcopy in Women With Cervical Dysplasia: a Randomized Controlled Trial.
Brief Title: LLETZ With Videocolposcopy Versus LLETZ With Binocular Colposcopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONE-5
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Uterine Cervical Dysplasia
Keywords: conization; LLETZ; randomized controlled trial; colposcopy; binocular colposcopy; intraoperative colposcopy; videocolposcopy; loop excision
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLETZ with videocolposcopy (Experimental): The LLETZ procedure will be performed using a videocolposcopy
  Interventions: Device: LLETZ with videocolposcope
- LLETZ with binocular colposcopy (Active Comparator): The LLETZ procedure will be performed using a binocular colposcope
  Interventions: Device: LLETZ with binocular colposcope

INTERVENTIONS:
Device: LLETZ with videocolposcope — Loop procedure using a videocolposcope in order to see and remove the abnormal cervical tissue
  Arms: LLETZ with videocolposcopy
Device: LLETZ with binocular colposcope — Loop procedure using a binocular colposcope in order to see and remove the abnormal cervical tissue
  Arms: LLETZ with binocular colposcopy

SUMMARY:
To assess the benefits of performing large Loop excision of the transformation Zone (LLETZ) using videocolposcopy compared to binocular colposcopy.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven cervical dysplasia
* colposcopy Prior to conization
* informed consent

Exclusion Criteria:

* significant language barrier
* a personal history of conization
* pregnancy
* the use of blood thinner
* unwillingness to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
the resected cone mass | 10 minutes
  the resected cone mass will be quantified by weighing the removed tissue with a precision scale located in the operating room

SECONDARY OUTCOMES:
Margin status | 2 Days after conization
  Resection margin is judge as "R0" if abnormal cells are not found in the margin of the biopsy or "R1" if abnormal cells remain in the margin of the biopsy. The histopathological examination will be done by an Independent pathologist
Operation time | 20 minutes
  the time from the beginning of the Operation (start of the electrosurgical method) until the end of the operation (the end of hemostatic interventions) will be measured in minutes
Operative complications | 14 days
  Operative complications defined as necessity to intervene therapeutically up to 14 days postoperatively
number of fragments of the surgical specimen | 10 minutes
  surgeons will count the number of the surgical specimen (1 vs. >1)
The circumference of the surgical specimens | 2 Days after conization
  The circumference of the surgical specimens will be measured in cm
the length of the surgical specimens | 2 Days after conization
  The length of The surgical specimens will be measured in cm
the thickness of the surgical specimens | 2 Days after conization
  The thickness of The surgical specimens will be measured in cm
handling of the device | 30 minutes
  surgeons will score their preference regarding the surgical method using an 11-step visual analogue scale (VAS) for ,(ranging from 0 (,very easy') to 10 (,very difficult')
satisfaction with the device | 30 minutes
  surgeons will score their preference regarding the surgical method using an 11-step visual analogue scale (VAS) for ,satisfaction with the device' (ranging from 0 (,very satisfied') to 10 (,absolutely not satisfied')
Time to complete intraoperative hemostasis | 120 seconds
  the time until complete hemostasis as judged by the surgeon has been achieved, will be measured in seconds
Intraoperative blood loss | 5 hours
  intraoperative blood loss will be measured using the difference in serum hemoglobin one day prior to surgery and within 5 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, M.D., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (1):
- Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezniczek GA, Neghabian N, Rehman S, Tempfer CB. Video colposcopy versus headlight for large loop excision of the transformation zone (LLETZ): a randomised trial. Arch Gynecol Obstet. 2022 Feb;305(2):415-423. doi: 10.1007/s00404-021-06331-0. Epub 2021 Nov 21. PMID 34802113